CLINICAL TRIAL: NCT04093609
Title: Detection of XIST Gene Deletion by Fluorescence in Situ Hybridization in Patients With Breast Cancer and Its Relation With Different Response to Therapies
Brief Title: XIST Gene Deletion in Breast Cancer Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, CN Fayez, principal investigator, Assiut University
Other Study IDs: Xist
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases
  Interventions: Genetic: XIST gene deletion
- control
  Interventions: Genetic: XIST gene deletion

INTERVENTIONS:
Genetic: XIST gene deletion — detection of XIST gene deletion by fluorescence in situ hybridization

SUMMARY:
Very little is known about the role of X-inactive specific transcript RNA in human breast cancer and in regulating different response to therapy .

the relation between the breast cancer predisposing gene BRCA1 & X-inactive specific transcript RNA has been investigated but still controversial.

Loss of X chromosome inactivation (XCI) is observed in breast cancer . Other studies sheds light on a possible mechanism of breast carcinogenesis mediated by XIST misbehaviour.

DETAILED DESCRIPTION:
breast cancer is an important cause of morbidity and mortality in women .Genetics of female contributes to her risk of having breast cancer . this disease is still discovered in their late stages due to the negligence of females inspite of self inspection and clinical examination of the breast .the identification of markers that could predict the tumor behavior is important in breast cancer management , staging, evaluation of therapeutic response and development of new therapeutic modalities .XIST (X-inactive specific transcript) RNA is a long non -coding RNA which plays an important role in inactivation of x_ chromosome which act as an example for long non _ coding RNA mediated gene regulation .Very little is known about the role of XIST in human breast cancer and in regulating different response on therapy . the relation between the breast cancer predisposing gene BRCA1 & XIST has been investigated but still controversial .Loss of X chromosome inactivation (XCI) is observed in breast . some studies provide evedience that BRCA1 Is involved in XIST regulation on the active X chromosome but not its localization .other studies sheds light on a possible mechanism of breast carcinogenesis mediated by XIST misbehaviour .

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients of breast cancer admitted to south egypt cancer institute at different stages of the disease

Exclusion Criteria:

* Other malignant diseases. Male breast cancer . Female with other sex linked diseases . Patients received chemotherapy for breast cancer .

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed female patients of breast cancer admitted to south egypt cancer institute above age of 20 years at different stages of the disease
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
detection of X inactive specific transcript RNA deletion in patients with breast cancer | 3 years
  detection of X inactive specific transcript RNA deletion by fluorescence in situ hybridization in patients with breast cancer and its relation with different response to therapies

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lima ZS, Ghadamzadeh M, Arashloo FT, Amjad G, Ebadi MR, Younesi L. Recent advances of therapeutic targets based on the molecular signature in breast cancer: genetic mutations and implications for current treatment paradigms. J Hematol Oncol. 2019 Apr 11;12(1):38. doi: 10.1186/s13045-019-0725-6. PMID 30975222
- [Background] Akram M, Iqbal M, Daniyal M, Khan AU. Awareness and current knowledge of breast cancer. Biol Res. 2017 Oct 2;50(1):33. doi: 10.1186/s40659-017-0140-9. PMID 28969709
- [Background] Yue M, Charles Richard JL, Yamada N, Ogawa A, Ogawa Y. Quick fluorescent in situ hybridization protocol for Xist RNA combined with immunofluorescence of histone modification in X-chromosome inactivation. J Vis Exp. 2014 Nov 26;(93):e52053. doi: 10.3791/52053. PMID 25489864
- [Background] Giudice A, Barbieri A, Bimonte S, Cascella M, Cuomo A, Crispo A, D'Arena G, Galdiero M, Della Pepa ME, Botti G, Caraglia M, Capunzo M, Arra C, Montella M. Dissecting the prevention of estrogen-dependent breast carcinogenesis through Nrf2-dependent and independent mechanisms. Onco Targets Ther. 2019 Jun 24;12:4937-4953. doi: 10.2147/OTT.S183192. eCollection 2019. PMID 31388303
- [Background] Banin Hirata BK, Oda JM, Losi Guembarovski R, Ariza CB, de Oliveira CE, Watanabe MA. Molecular markers for breast cancer: prediction on tumor behavior. Dis Markers. 2014;2014:513158. doi: 10.1155/2014/513158. Epub 2014 Jan 28. PMID 24591761